CLINICAL TRIAL: NCT06525584
Title: Ketamine Infusion in the Postoperative Period as a Method of Cerebral Protection in Children During Surgical Correction of Congenital Heart Defects
Brief Title: Ketamine Infusion as a Method of Cerebral Protection in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kemerovo State Medical University (Other)
Responsible Party: Principal Investigator, Evgeny Grigoryev, Head of the Department of Anesthesiology, Kemerovo State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketamine 1 (Experimental)
  Interventions: Drug: Ketamine Hcl 50Mg/Ml Inj
- Ketamine 3 (Experimental)
  Interventions: Drug: Ketamine Hcl 50Mg/Ml Inj
- Control (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Drug: Ketamine Hcl 50Mg/Ml Inj — ketamine infusion at a dose of 0.1 mg/kg/hour for 16 hours
  Arms: Ketamine 1
Drug: Ketamine Hcl 50Mg/Ml Inj — ketamine infusion at a dose of 0.3 mg/kg/hour for 16 hours
  Arms: Ketamine 3
Other: Control — Without ketamine
  Arms: Control

SUMMARY:
The study is devoted to the use of ketamine infusion in a subanesthetic dose in the postoperative period in children after surgical correction of congenital heart defects in children.

DETAILED DESCRIPTION:
The study will examine the safety and effectiveness for neuroprotection of subanesthetic doses of ketamine in the postoperative period in children undergoing operations to correct septal congenital heart defects using cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* age from 1 to 60 months
* body weight from 3.5 to 20 kg
* planned surgical intervention to correct a congenital heart defect (atrial or ventricular septal defect) with CPBё
* the presence of informed consent for participation in the study signed by the child's legal representative

Exclusion Criteria:

* lack of informed consent of the patient and parents to participate in the study,
* emergency and urgent surgical interventions;
* the presence of clinically significant anemia;
* hypo-thermic during operation, episodes of desaturation in the perioperative period;
* the presence of another congenital heart diseases besides the atrial or ventricular septal defect, as well as their combination;
* a history of central nervous system diseases;
* an installed pacemaker;
* hemodynamic instability requiring preoperative pharmacological and/or mechanical support;
* any episodes of cerebrovascular accidents in the history or periop-erative period;
* the presence of a patient with severe concomitant diseases that worsen mental and somatic conditio;
* acute infection and exacerbation of chronic infection in the perioperative period;
* concomitant autoimmune diseases;
* the presence of malignant neoplasms;
* surgical complications in the postoperative period.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers | 16 hours after operation
  monitoring the concentration of markers of brain damage at several control points

CONTACTS AND LOCATIONS:
Locations (1):
- Artem Ivkin, Kemerovo, Please Select, Russia

IPD SHARING:
Plan to Share IPD: No